CLINICAL TRIAL: NCT02423707
Title: Intralymphatic Allergen-specific Immunity as a New Administration Route for Treatment of Pollen-induced Allergic Diseases
Brief Title: Safety and Efficacy Study of Intralymphatic Allergen-specific Immunotherapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Skane University Hospital (Other); Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Lars Olaf Cardell, Professor, Head of Division, MD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-016815-39
Record Dates: First submitted 2012-03-28; First posted 2015-04-22 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALK Alutard Birch and/or 5-grasses (Active Comparator): 3 intralymphatic injections with dose 1000 SQ-U and dose interval 4 weeks.
  Interventions: Drug: ALK Alutard Birch and/or 5-grasses
- ALK diluent (Placebo Comparator): 3 intralymphatic injections with dose interval 4 weeks.
  Interventions: Drug: ALK Diluent

INTERVENTIONS:
Drug: ALK Alutard Birch and/or 5-grasses — 3 intralymphatic injections of 1000 SQ-U birch and/or grass allergen with 4 weeks interval.
  The substance used for the three intralymphatic injections is ALK-alutard SQ Betula verrucosa® and ALK-alutard SQ 5-grasses ® under ATC-code V01AA, V04CL and V07AB which is a depot formulation for subcutaneous use.
  Other Names: ALK Alutard Betula Verrucosa and ALK Alutard 5-grasses
  Arms: ALK Alutard Birch and/or 5-grasses
Drug: ALK Diluent — This placebo group will receive 3 injections of 0.3% human albumin instead of active substance
  Other Names: Human albumin
  Arms: ALK diluent

SUMMARY:
Allergen-specific immunotherapy (ASIT) is commonly used to treat patients with allergic rhino-conjunctivitis and asthma, and it is the only proven treatment that affects the long-term development of allergic rhinitis and asthma. The current treatment regime of ASIT requires numerous subcutaneous allergen injections and takes several years to complete. Hence, there is a need to develop more convenient protocols for induction of allergen tolerance.

Emerging evidence suggest that by targeting of antigen presenting cells within the lymph nodes the immunogenicity of the allergen can be enhanced and the number of injections can be reduced.

The purpose of this study is to evaluate whether intralymphatic administration of ASIT is a safe and effective treatment for patients with pollen-induced allergic rhinitis. The long term goal is to provide a base for a more efficient administration of ASIT, which will reduce both the dose necessary and the number of clinic visits associated with the conventional subcutaneous ASIT.

The investigators will make an attempt to reproduce the results of a recent human study of intralymphatic ASIT (clinicaltrials.gov; NCT00470457) in a Swedish clinical setting.

The first part of the study is completed and published (PMID: 23374268)

DETAILED DESCRIPTION:
In the first part of the study safety and clinical efficacy of ALK Alutard Birch or 5-grass have been evaluated in a RCT with 50 patients. Active patients recieve 3 injections with 1000 SQ-U ALK Alutard or 5-grasses in a lymph node in the groin. Dose interval 4 weeks. This part of the study is completed and published (PMID: 23374268)

In the second part of the study 60 patients participates in a RCT with intralymphatic injections with both ALK Alutard Birch AND ALK Alutard 5-grasses. The injections are given intralymphatically with one allergen in each groin with 30 minutes observation between injections. Dose and dose interval are the same as in the first part of the study; the active group recieves 1000 SQ-U ALK Alutard Birch in right groin and 1000 SQ-U 5-grasses in left groin. The injections are given 3 times with 4 weeks interval. Enrollment and treatment is completed and the results will be evaluated in the autumn 2015.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50,
* Seasonal allergic symptoms for birch and/or grass verified by skin prick test,
* Accepted informed consent

Exclusion Criteria:

* Pregnancy or nursing
* Autoimmune or collagen disease (known)
* Cardiovascular disease
* Perennial pulmonary disease
* Hepatic disease
* Renal disease
* Cancer
* Any medication with a possible side-effect of interfering with the immune response
* Previous immuno- or chemotherapy
* Chronic diseases
* Other upper airway disease (non-allergic sinusitis, nasal polyps, chronic obstructive and restrictive lung disease)
* Disease or conditions rendering the treatment of anaphylactic reactions difficult (symptomatic coronary heart diseases, severe arterial hypertension and treatment with β-blockers)
* Major metabolic disease
* Known or suspected allergy to the study product
* Alcohol or drug abuse
* Mental incapability of coping with the study
* Withdrawal of informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2010-08; Primary Completion 2015-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in subjective allergic symptoms following nasal allergen provocation | Before treatment, an average of 4 weeks after completed treatment and 6-9 months after treatment.
  The study subjects will be intranasally challenged with allergen and symptom score questionnaires are filled out pre-provocation and 5, 10 and 30 min post-provocation.

SECONDARY OUTCOMES:
Registration of adverse event | from the first injection to 30 days after the last injections has been given
Effects on quality of life | During peak pollen season which will be up to 5 months (birch) and 6 months (grass) after completed treatment
  SNOT-22 questionnaire
Effects on quality of life | During peak pollen season which will be up to 5 months (birch) and 6 months (grass) after completed treatment
  Juniper RQLQ questionnaires
Change in medicine consumption during pollen season | 6-9 months after treatment.
  After the pollen season patients report to what extension they have been using medications; more, the same or less. The mediacations asked about are antihistamine tablets, antihistamine eye drops, nasal steroid, steroid tablets, b2-bronchodilator inhalation, leucotrien receptor antagonist, nasal or ocular sodium chromoglycates.
Change in symptoms at pollen season | 6-9 months after treatment.
  After the pollen season at the 6-9 months follow up patients recall the pollen season and rates the improvement on an arbitrary scale ranging 0-10 with 0 as "no improvement at all" and 10 "total symptom relief".
Short term improvement of skin reactivity | Before treatment, an average of 4 weeks after completed treatment and 6-9 months after treatment.
  Skin prick test
S-IgE Birch | Before treatment, approximately 4 weeks after completed treatment and 6-9 months after treatment
S-IgE Grass | Before treatment, approximately 4 weeks after completed treatment and 6-9 months after treatment
S-IgG4 Grass | Before treatment, approximately 4 weeks after completed treatment and 6-9 months after treatment
S-IgG4 Birch | Before treatment, approximately 4 weeks after completed treatment and 6-9 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Olaf Cardell, Prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Allergic Unit at the Department of Oto-Rhino-Laryngology at Skåne University Hospital Malmö, Malmo, Sweden

REFERENCES:
- [Background] Senti G, Prinz Vavricka BM, Erdmann I, Diaz MI, Markus R, McCormack SJ, Simard JJ, Wuthrich B, Crameri R, Graf N, Johansen P, Kundig TM. Intralymphatic allergen administration renders specific immunotherapy faster and safer: a randomized controlled trial. Proc Natl Acad Sci U S A. 2008 Nov 18;105(46):17908-12. doi: 10.1073/pnas.0803725105. Epub 2008 Nov 10. PMID 19001265